CLINICAL TRIAL: NCT05091554
Title: Effect of Intraoral Cryotherapy Application on Postoperative Pain in Nonsurgical Endodontic Retreatment of Teeth With Apical Periodontitis: A Randomized Clinical Trial
Brief Title: Intraoral Cryotherapy in Root Canal Retreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, emrah karataslioglu, Assoc. Prof. Dr., Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IzmirKCUekarataslioglu
Record Dates: First submitted 2021-09-28; First posted 2021-10-25 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Cryotherapy Effect
Keywords: analgesic; cryotherapy; periapical periodontitis; postoperative pain; retreatment
MeSH Terms: conditions — Periapical Periodontitis; Pain, Postoperative

STUDY DESIGN:
Masking Description: In this study, double blindness was not possible because of the nature of the ice packs, the patients and the physician were aware of the cryotherapy groups. Therefore, patients were only blinded before the treatment procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Single visit control (No Intervention): The root canals were obturated in the same session using cold lateral compaction technique with AH Plus sealer (Dentsply DeTrey, Konstanz, Germany), Protaper Universal gutta-percha (ProTaper Universal gutta-percha, Dentsply) and .02 tapered auxiliary gutta-percha (Diadent, Chongju, Korea) cones. Residual gutta-perchas in the access cavity were removed with the aid of heated hand tools. The quality of root canal filling was checked with periapical radiographs.
  The pulp chamber was filled with flowable composite resin (Filtek Ultimate Flowable, 3M-ESPE, St. Paul, MN, USA) and nanohybrid composite resin (3M-ESPE) using an incremental technique.
  Intraoral cryotherapy was not applied.
- Single visit 15 minutes cryotherapy (Experimental): The root canals were obturated in the same session using cold lateral compaction technique with AH Plus sealer (Dentsply DeTrey, Konstanz, Germany), Protaper Universal gutta-percha (ProTaper Universal gutta-percha, Dentsply) and .02 tapered auxiliary gutta-percha (Diadent, Chongju, Korea) cones. Residual gutta-perchas in the access cavity were removed with the aid of heated hand tools. The quality of root canal filling was checked with periapical radiographs.
  The pulp chamber was filled with flowable composite resin (Filtek Ultimate Flowable, 3M-ESPE, St. Paul, MN, USA) and nanohybrid composite resin (3M-ESPE) using an incremental technique.
  15 minutes intraoral cryotherapy was applied.
  Interventions: Procedure: intraoral ice pack application
- Single visit 30 minutes cryotherapy (Experimental): The root canals were obturated in the same session using cold lateral compaction technique with AH Plus sealer (Dentsply DeTrey, Konstanz, Germany), Protaper Universal gutta-percha (ProTaper Universal gutta-percha, Dentsply) and .02 tapered auxiliary gutta-percha (Diadent, Chongju, Korea) cones. Residual gutta-perchas in the access cavity were removed with the aid of heated hand tools. The quality of root canal filling was checked with periapical radiographs.
  The pulp chamber was filled with flowable composite resin (Filtek Ultimate Flowable, 3M-ESPE, St. Paul, MN, USA) and nanohybrid composite resin (3M-ESPE) using an incremental technique.
  30 minutes intraoral cryotherapy was applied.
  Interventions: Procedure: intraoral ice pack application
- Multiple visit control (No Intervention): Root canals were filled with calcium hydroxide paste (Kalsin, Turkey), prepared according to the rate recommended by the manufacturer using a lentulo spiral (Dentsply Sirona, Switzerland) 2 mm from the working length. Sterile dry cotton pellets were placed in the pulp chamber, then the access cavity was sealed with a temporary filling material and occlusion was checked.
  Intraoral cryotherapy was not applied. Patients were given an appointment 7 days later for second visit. In this appointment, patients were anesthetized, the tooth was isolated with rubber dam, the temporary filling material was removed. Then calcium hydroxide paste was removed by using the last instrument used to prepare the root canals at the working length during the first appointment using sufficient irrigation.
  The final irrigation protocol was repeated. Root canal fillings and permanent restorations were completed by applying the same techniques as in single session groups.
- Multiple visit 15 minutes cryotherapy (Experimental): Root canals were filled with calcium hydroxide paste (Kalsin, Turkey), prepared according to the rate recommended by the manufacturer using a lentulo spiral (Dentsply Sirona, Switzerland) 2 mm from the working length. Sterile dry cotton pellets were placed in the pulp chamber, then the access cavity was sealed with a temporary filling material and occlusion was checked.
  15 minutes intraoral cryotherapy was applied. Patients were given an appointment 7 days later for second visit. In this appointment, patients were anesthetized, the tooth was isolated with rubber dam, the temporary filling material was removed. Then calcium hydroxide paste was removed by using the last instrument used to prepare the root canals at the working length during the first appointment using sufficient irrigation.
  The final irrigation protocol was repeated. Root canal fillings and permanent restorations were completed by applying the same techniques as in single session groups.
  Interventions: Procedure: intraoral ice pack application
- Multiple visit 30 minutes cryotherapy (Experimental): Root canals were filled with calcium hydroxide paste (Kalsin, Turkey), prepared according to the rate recommended by the manufacturer using a lentulo spiral (Dentsply Sirona, Switzerland) 2 mm from the working length. Sterile dry cotton pellets were placed in the pulp chamber, then the access cavity was sealed with a temporary filling material and occlusion was checked.
  30 minutes intraoral cryotherapy was applied. Patients were given an appointment 7 days later for second visit. In this appointment, patients were anesthetized, the tooth was isolated with rubber dam, the temporary filling material was removed. Then calcium hydroxide paste was removed by using the last instrument used to prepare the root canals at the working length during the first appointment using sufficient irrigation.
  The final irrigation protocol was repeated. Root canal fillings and permanent restorations were completed by applying the same techniques as in single session groups.
  Interventions: Procedure: intraoral ice pack application

INTERVENTIONS:
Procedure: intraoral ice pack application — Tap water was filled into plastic ice molds and kept in the freezer in the clinic until the application was made. The ice packs used were weighed with digital pocket scale (Knmaster CT1000, Turkey) as 6-8 grams. In the cryotherapy groups, at the end of the first appointment ice packs were removed from the freezer, wrapped in sterile gauze and placed on the vestibular mucosa of the teeth.
  Arms: Multiple visit 15 minutes cryotherapy; Multiple visit 30 minutes cryotherapy; Single visit 15 minutes cryotherapy; Single visit 30 minutes cryotherapy

SUMMARY:
The aim of this study was to evaluate the effect of intraoral cryotherapy application on postoperative pain in single and multiple visit retreatment of teeth with symptomatic or asymptomatic apical periodontitis. This clinical trial was also investigate the potential of intraoral cryotherapy application to reduce on postoperative analgesic use of patients in line with the results obtained.

A total of 118 patients who met the inclusion criteria were selected for the study. The patients were randomly divided into two groups as single visit and multiple visit (n=59). Then, each group was randomly divided into three subgroups as control (without cryotherapy), 15 minutes of cryotherapy, and 30 minutes of cryotherapy. Twenty two teeth were retreated in each cryotherapy group and 15 teeth in each control group. Visual analogue scale (VAS) was used to evaluate and compare postoperative pain. Postoperative analgesic use of patients was also recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 65 year-old patients.
* Patients with pre-treated teeth diagnosed with symptomatic or asymptomatic apical periodontitis.
* Patients who can tolerate the treatment physically and mentally.

Exclusion Criteria:

* The presence of any systemic disease,
* the presence of any allergic reactions or pregnancy,
* use of any analgesic or antibiotic medication within 7 days,
* use of corticosteroid within 6 months,
* severe periodontal disease (periodontal pockets >3 mm) in the pretreated tooth,
* surgical endodontic treatment,
* having drainage,
* periapical index (PAI) score 1 and 2,
* excessively curved, excessively long or short roots, calcified or resorbed root canals,
* immature apices,
* complications like perforation, overfilling, broken files

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2020-03-14 (Actual)

PRIMARY OUTCOMES:
Levels of postoperative pain | 6 hours
  The primary endpoint in calculating the sample size was to obtain visual analog scale (VAS) values. The intensity of postoperative pain was evaluated with visual analogue scale, which is a 10 cm line representing a continuum of pain levels between "no pain" on the left side and "most severe pain" on the right side between 0 and 10.
Levels of postoperative pain | 24 hours
  The primary endpoint in calculating the sample size was to obtain visual analog scale (VAS) values. The intensity of postoperative pain was evaluated with visual analogue scale, which is a 10 cm line representing a continuum of pain levels between "no pain" on the left side and "most severe pain" on the right side between 0 and 10.
Levels of postoperative pain | 72 hours
  The primary endpoint in calculating the sample size was to obtain visual analog scale (VAS) values. The intensity of postoperative pain was evaluated with visual analogue scale, which is a 10 cm line representing a continuum of pain levels between "no pain" on the left side and "most severe pain" on the right side between 0 and 10.
Levels of postoperative pain | 1 week
  The primary endpoint in calculating the sample size was to obtain visual analog scale (VAS) values. The intensity of postoperative pain was evaluated with visual analogue scale, which is a 10 cm line representing a continuum of pain levels between "no pain" on the left side and "most severe pain" on the right side between 0 and 10.

SECONDARY OUTCOMES:
Rate of analgesic use | 1 week
  Comparison of analgesic use in groups

CONTACTS AND LOCATIONS:
Overall Officials: emrah karataslioglu, phd, Principal Investigator — Izmir Katip Celebi University; sule soysal, DDS, Principal Investigator — Izmir Katip Celebi University; ılgın akçay, phd, Principal Investigator — Ege University
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)